CLINICAL TRIAL: NCT00409279
Title: An Innovative Psychosocial Intervention for Adult-Child Caregivers of Parents With Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Jacob and Valeria Langeloth Foundation (Other)
Responsible Party: Joseph E. Gaugler, Ph.D., Assistant Professor, University of Minnesota, School of Nursing
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IA0097; Project #195
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Alzheimer Disease
Keywords: Aging; Parent / Adult-child interaction; Family caregivers; Alzheimer's; Caregiving
MeSH Terms: conditions — Alzheimer Disease | interventions — Counseling; Palliative Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): multi-component psychosocial intervention
  Interventions: Behavioral: Information, counseling and support
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Information, counseling and support — individual-family consultation, support group, and ad hoc consultation
  Arms: 1

SUMMARY:
The goal of this project is to test an intervention designed to reduce the incidence and magnitude of the negative effects, specifically stress, anxiety, and depression, frequently experienced by adult children who are caregivers of a parent with Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Caring for an elderly parent is a growing societal problem, and many studies have shown that caring for a person with dementia can have a negative impact on a caregiver's psychological and physical health, social life and career, and relationship with the patient. Stress and coping models proposed in the AD caregiving literature, and general stress and coping theories suggest that by improving caregivers' ability to cope and master the caregiving situation, it is possible to avoid or ameliorate the negative emotional consequences of caregiving.

Building upon the results of a pilot study, this study will formally test the efficacy of a psychosocial intervention, based on a concept of caregiving that builds on the interests, activities, and responsibilities of both the caregiver and patient in creating a care strategy. The intervention is designed to reduce the negative effects frequently experienced by adult children who care for a parent in the middle stage of Alzheimer's disease. Caregivers will learn to engage with their parents in activities that are within the patients' remaining functional and cognitive abilities. Caregivers will also be encouraged to teach activities to other family members and paid caregivers. The study will also evaluate a lower level of intervention, based on written materials.

It is expected that by increasing knowledge about AD and providing what may be a new conceptual approach to relating to a parent at this point in the disease process, 1) caregivers and patients may experience a higher level of satisfaction and gratification from their interactions, 2) caregivers will gain a sense of control and mastery over a difficult situation and thus feel more capable of coping and 3) the patient may maintain a higher level of functioning.

A randomized treatment/control design will be used, and adult-child caregivers who participate will be assigned to one of the two levels of intervention, each designed to reduce stress, anxiety and depression. The benefits of each intervention will be evaluated by looking at the change in scores on widely used measures of the anticipated outcomes among caregivers in each group, and their relative benefits will be tested by comparing scores of the caregivers in the two groups at two follow-up points, six and nine months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 21 and 90
* Adult-child caring for at least one parent who has been diagnosed with Alzheimer's disease and is in the moderate stage
* Person with Alzheimer's disease must be living at home or in a congregate residential setting that is like a home
* Caregiver must be willing to complete intake and follow-up questionnaires
* Caregiver must be willing to attend 2 workshops and 1 individual counseling session

Exclusion Criteria:

* Severe psychological or physical illness
* Unwillingness to participate in all aspects of the study

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-09; Primary Completion 2008-04 (Estimated); Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
Changes in measures of depression, stress, and anxiety | six and nine months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mary S. Mittelman, DrPH, Principal Investigator — NYU School of Medicine
Locations (1):
- Aging and Dementia Research Center, Silberstein Institute, NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Mittelman MS, Ferris SH, Shulman E, Steinberg G, Ambinder A, Mackell JA, Cohen J. A comprehensive support program: effect on depression in spouse-caregivers of AD patients. Gerontologist. 1995 Dec;35(6):792-802. doi: 10.1093/geront/35.6.792. PMID 8557206
- [Background] Mittelman MS, Ferris SH, Shulman E, Steinberg G, Levin B. A family intervention to delay nursing home placement of patients with Alzheimer disease. A randomized controlled trial. JAMA. 1996 Dec 4;276(21):1725-31. PMID 8940320